CLINICAL TRIAL: NCT00400036
Title: Assessment of Insulin Sensitivity in Insulin-Resistant Subjects Fed Fish Protein
Brief Title: Dietary Fish Protein in Subjects With Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MOP-64443
Record Dates: First submitted 2006-11-14; First posted 2006-11-16 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2006-11

CONDITIONS: Insulin Resistance; Type 2 Diabetes
Keywords: cod protein; insulin sensitivity; plasma lipids; glucose tolerance; plasma inflammatory markers; skeletal muscle insulin signaling; type 2 diabetes; humans
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: Cod protein NCEP-diet

SUMMARY:
The objective of our research project is to determine the effects of fish protein, present in fish, on insulin sensitivity in insulin-resistant human individuals, and its mechanism of action on glucose metabolism. Our hypothesis is that fish protein improves insulin sensitivity, glucose tolerance and plasma lipid profile through an improvement in a primary defect in insulin signaling in overweight and insulin-resistant subjects.

DETAILED DESCRIPTION:
Recent data show that cod protein prevents the development of insulin resistance in rats. Dietary fish protein may also enhance insulin sensitivity in overweight insulin-resistant subjects by improving a primary defect in insulin signaling to PI 3-kinase, leading to reduced activation of the downstream effectors Akt and PKC. To determine whether this is the case, we will study the effects of fish protein on insulin sensitivity in humans, and how it improves the ability of muscles to use glucose. Such studies will help to advise individuals with insulin resistance or type 2 diabetes about eating fish.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (BMI between 25 and 40 kg /m2)
* waist circumference above 88 cm for women and 102 cm for men
* fasting plasma insulin above 90 pmol/L
* fasting plasma glucose below 7.0 mmol/L and 2-h plasma glucose below 11.1 mmol/L

Exclusion Criteria:

* Individuals with diagnosed diabetes or any chronic, metabolic or acute disease
* Individuals who had a major surgery within the last 3 months
* Individuals who had a significant weight loss (±10%) within the last 6 months
* Individuals taking any medication known to affect lipid or glucose metabolism
* Subjects with dietary incompatibility with fish consumption (allergy, intolerance or dislike) and/or calcium supplementation
* Smokers

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-02; Study Completion 2005-12

PRIMARY OUTCOMES:
Insulin sensitivity at 4 weeks
Insulin signaling in skeletal muscle at 4 weeks

SECONDARY OUTCOMES:
plasma lipids and lipoproteins at 4 weeks
plasma inflammatory markers at 4 weeks
glucose tolerance at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helene Jacques, PhD, Principal Investigator — Laval University; Andre Marette, PhD, Principal Investigator — Laval University; Stanley J Weisnagel, MD / FRCPC, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Ouellet V, Marois J, Weisnagel SJ, Jacques H. Dietary cod protein improves insulin sensitivity in insulin-resistant men and women: a randomized controlled trial. Diabetes Care. 2007 Nov;30(11):2816-21. doi: 10.2337/dc07-0273. Epub 2007 Aug 6. PMID 17682120